CLINICAL TRIAL: NCT06226233
Title: Efficacy of Juniver, a Digital Self-help Intervention, on Symptoms of Eating Disorders: A Randomised Controlled Trial
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: Juniver (Industry); Innovate UK (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JUNIVER-ED001; HR/DP-23/24-39714 (Other: King's College London Research Ethics Committee); 10060885 (Other Grant/Funding Number: Innovate UK)
Record Dates: First submitted 2024-01-17; First posted 2024-01-26 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-03

CONDITIONS: Feeding and Eating Disorders; Anorexia Nervosa; Bulimia Nervosa; Binge-Eating Disorder; Binge Eating; Eating Disorders; Disordered Eating
Keywords: Eating disorders; Anorexia nervosa; Bulimia nervosa; Binge eating disorder; Just in time interventions; Digital interventions; Mental health
MeSH Terms: conditions — Feeding and Eating Disorders; Anorexia Nervosa; Bulimia Nervosa; Binge-Eating Disorder; Bulimia; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: The Juniver program is a self-help intervention for eating disorders delivered digitally, through an iPhone app. It features three components: an evidence-based curriculum, interactive tools, and moderated peer support groups. This trial aims to investigate the impact of the Juniver program on self-reported eating disorder symptoms, as well as on symptoms of depression, anxiety, psychosocial impairment associated with eating disorders, and perceived stress. This will occur via a randomised controlled trial comparing Juniver to a wait-list control condition over a 12-week period, with further evaluation of the effects of Juniver up to 24-weeks.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Juniver intervention group (Experimental): Immediate access to the Juniver program
  Interventions: Other: Juniver program
- Wait list control (No Intervention): Access to the Juniver program after 12 weeks

INTERVENTIONS:
Other: Juniver program — The Juniver program is a self-help intervention for eating disorders delivered digitally, through an iPhone app. It features three components: an evidence-based curriculum, interactive tools, and moderated peer support groups.
  Arms: Juniver intervention group

SUMMARY:
This project aims to assess the efficacy of the Juniver program on symptoms of eating disorders via a randomised controlled trial. The Juniver program is a self-help intervention for eating disorders delivered digitally, through an iPhone app. It features three components: an evidence-based curriculum, interactive tools, and moderated peer support groups.

These three components integrate the evidence for (a) Cognitive-Behavioural Therapy (CBT) and Dialectical Behaviour Therapy for eating disorders; (b) Just-in-Time Adaptive Intervention; and (c) peer mentorship as an adjunct intervention for the treatment of eating disorders.

The program was developed by the Juniver team made up of people with lived experience with eating disorders and professional experience in digital health, a panel of neuroscientists and experts specialising in eating disorders, and direct research with 500 participants.

This trial aims to investigate the impact of the Juniver program on self-reported eating disorder symptoms, as well as on symptoms of depression, anxiety, psychosocial impairment associated with eating disorders, and perceived stress. This will occur via a randomised controlled trial comparing Juniver to a wait-list control condition over a 12-week period, with further evaluation of the effects of Juniver up to 24-weeks.

DETAILED DESCRIPTION:
Background Eating disorders are psychiatric disorders defined by extreme and life-threatening behaviours surrounding weight and food intake. Every year, eating disorders affect 2.4m people in the UK, costing £12bn, and 28.8m in the US, costing $65b (Beat, 2015; Deloitte Access Economics, 2020; The Hearts Minds and Genes Coalition for Eating Disorders, 2021). The problem is growing: hospitalisations for eating disorders are up 84% and over half of female university students report some symptoms of an eating disorder. Symptoms are very disruptive and eating disorders are associated with significant and persistent impairments in quality of life. Medical costs for those with eating disorders are up to 7.2x higher than those without behavioural health conditions (Beat, 2015).

Current treatments for eating disorders are moderately effective at best, and, on average, only 1 in 4 individuals with eating disorders access specialist help for their condition (Ali et al., 2017; Hart et al., 2011). While women represent the majority of sufferers, eating disorders affect people of any weight, age, gender, socioeconomic background and ethnicity (Beat, 2015). Yet, less than a third of published papers reflect that diversity, fuelling the stereotype of the typical sufferer being an underweight, White young woman.

The sector is ripe for innovation, especially today when technological tools can serve clinical needs, and the vast majority of the UK & US population has a smartphone in their pocket. Juniver Limited collaborated with leading clinicians and hundreds of sufferers including underserved groups to establish what could be done better. We found that all eating disorders are characterised by urges, and that the moment of experiencing an urge is when help is most needed and impactful. Overcoming an urge paves the way to recovery by decreasing the intensity and frequency of subsequent urges - this is how most smokers quit smoking, for example. It's particularly difficult for eating disorder sufferers to overcome urges unsupported, as they have to eat for sustenance and are triggered multiple times every day. We developed a solution rooted in the science of addiction that delivers micro-interventions for on-demand help in compulsive moments (Baumel, Fleming & Schueller, 2020; Johnson et al., 2022; Juarascio et al., 2018).

A pilot with 97 users validated demand and engagement, with strong signals that our solution works (92% of those who tried our main tool successfully overcame an urge). Additionally, we conducted direct research with 500 participants. We uncovered the following:

* Sufferers are desperate to get better: 97% have sought treatment before, in most (92%) cases, unsuccessfully.
* When asked why they haven't yet recovered, 73% 'haven't found something that's worked' or 'don't know how to recover.'
* The top 3 barriers to access are cost, stigma, and the complexity of navigating specialist care systems.

The Juniver program was developed to directly address these findings. This clinical trial will help advance understanding of how Juniver works and for whom, allow for research with a more diverse population of individuals than those presenting to clinical services, and inform the ways self-guided, on-demand help can contribute to better, more equitable outcomes.

Clinical trial The study will include a sample of 300 participants aged 16 years and over, with participants randomly allocated at a 1:1 ratio to the immediate Juniver group (n=150) or wait-list control group (n=150). The total sample size of 300 participants was guided by statistical power calculations performed using G*Power 3 software. This factors in a drop-off rate of 30%, estimated from similar studies involving digital interventions for eating disorders and other mental health disorders. Participants assigned to the Juniver group will gain access to the app starting on their respective Week 1. In contrast, participants in the control group will receive access to the app at the conclusion of their respective Week 12. The Juniver group will complete outcome measures at Week 4, 8, 12, 16, 20 and 24 while the control group will complete measures at Week 4, 8 and 12. Statistical analysis will involve linear mixed models to compare differences in outcome measures in the Juniver group compared to the control group, including any overall between-group differences and any differences in how variables change over time.

ELIGIBILITY:
Inclusion Criteria:

* Aged 16 or over
* Live in the UK or the US
* Any presence and severity of any eating disorder(s): Anorexia Nervosa, Bulimia Nervosa, Binge Eating Disorder, Other Specified Feeding and Eating Disorders (OSFED), Avoidant Restrictive Food Intake Disorder (ARFID) and Unspecified Feeding or Eating Disorder (UFED) as measured by the EDE-Q and using item-based algorithms to determine the potential presence of one of these eating disorders
* Able to provide informed consent
* Willing to provide full contact details including a UK or US address, phone number and email address
* Willing to provide contact details for a health care professional with whom they are registered (e.g., a general practitioner or primary care physician) and who the study team can contact if they are concerned about their well-being.

Exclusion Criteria:

* Lack of access to an iPhone - as Juniver is currently only available for use on the iPhone system.
* Partaking in any medically-driven special diets (e.g., linked to Coeliac, Crohn's, PCOS, type 1 or type 2 diabetes) - as these individuals would require more specialist dietary advice than the Juniver program can safely provide. Individuals with these conditions who are not on special diets would be eligible to enrol.
* Severe depression as measured by PHQ score > 20
* Active suicidal intent or plan

  .- Body Mass Index (BMI) <15
* Emergency hospital visit or admission within the last month for an eating disorder or other mental health concern

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-12-23 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Eating Disorder Examination-Questionnaire (EDE-Q) Eating Disorder Examination-Questionnaire (EDE-Q) | 12 weeks
  Self-report measure of eating disorder symptoms

SECONDARY OUTCOMES:
Patient Health Questionnaire-9 (PHQ-9) | 12 weeks
  Self-report measure of depressive symptoms
Generalised Anxiety Disorder-7 questionnaire (GAD-7) | 12 weeks
  Self-report measure of anxiety symptoms
Clinical Impairment Questionnaire (CIA 3.0) | 12 weeks
  Self-report measure of psychosocial impairment due to an eating disorder
Perceived Stress Scale (PSS-4) | 12 weeks
  Self-report measure of perceived stress

OTHER OUTCOMES:
Acceptability of the Juniver program | 24 weeks
  Net Promoter Score (how likely are you to recommend the Juniver app to others) from 0-10

CONTACTS AND LOCATIONS:
Overall Officials: Karina Allen, PhD, Principal Investigator — King's College London
Locations (1):
- King's College London, London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No data sharing planned

REFERENCES:
- See also: Trial website — https://www.junivertrial.com/